CLINICAL TRIAL: NCT07360353
Title: A Comparative Study of Performance and Cost-effectiveness of Three Different Single-Use Flexible Ureteroscopes in the Management of Renal Stones: A Randomized Clinical Trial
Brief Title: Comparison Between Different Types of Flexible Ureteroscopes
Acronym: FURS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hesham Elsayed Mohammed, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 788/2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Renal Calculi; Nephrolithiasis
Keywords: Flexible ureteroscopy; Single-use flexible ureteroscope; Renal stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LithoVue™ (Boston Scientific Corporation) (Active Comparator): Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the LithoVue™ single-use digital flexible ureteroscope.
  Interventions: Device: LithoVue™ (Boston Scientific Corporation)
- WiScope® (OTU Medical Inc. (Silicon Valley, USA)) (Active Comparator): Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the WiScope® single-use digital flexible ureteroscope.
  Interventions: Device: WiScope® (OTU Medical Inc. (Silicon Valley, USA))
- Single-Use Ureterorenoscope (Scivita Medical Technology Co., Ltd.) (Active Comparator): Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the single-use digital flexible ureterorenoscope manufactured by Scivita Medical Technology Co., Ltd.
  Interventions: Device: Single-Use Ureterorenoscope (Scivita Medical Technology Co., Ltd.)

INTERVENTIONS:
Device: LithoVue™ (Boston Scientific Corporation) — Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the LithoVue™ single-use digital flexible ureteroscope.
  Arms: LithoVue™ (Boston Scientific Corporation)
Device: WiScope® (OTU Medical Inc. (Silicon Valley, USA)) — Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the WiScope single-use digital flexible ureteroscope.
  Arms: WiScope® (OTU Medical Inc. (Silicon Valley, USA))
Device: Single-Use Ureterorenoscope (Scivita Medical Technology Co., Ltd.) — Participants randomized to this arm will undergo retrograde intrarenal surgery (RIRS) for renal stone management using the single-use digital flexible ureterorenoscope manufactured by Scivita Medical Technology Co., Ltd.
  Arms: Single-Use Ureterorenoscope (Scivita Medical Technology Co., Ltd.)

SUMMARY:
The current study aims to compare the performance of three distinct single-use digital flexible ureteroscope types in terms of cost-effectiveness, postoperative complications, operating time, and stone-free rates (SFRs).

DETAILED DESCRIPTION:
Retrograde intrarenal surgery (RIRS) is the preferred treatment modality for renal stones measuring less than 20 millimeters (mm). Several types of flexible ureteroscopes are currently available on the market from different manufacturers. However, there is a shortage of comparative studies evaluating the performance of different single-use flexible ureteroscopes.

This study aims to compare the performance of three different single-use digital flexible ureteroscopes in terms of cost-effectiveness, postoperative complications, operative time, and stone-free rates (SFRs).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 years.
* Presence of renal stones measuring less than 20 millimeters (mm).

Exclusion Criteria:

* Renal stones larger than 20 millimeters (mm).
* Uncontrolled bleeding disorders or coagulopathies.
* Active urinary tract infection.
* Renal failure.
* Uncontrolled diabetes mellitus, hypertension, or hepatic dysfunction.
* Pregnancy.
* Abnormal urinary tract anatomy or known ureteric stricture.
* History of previous open ureteric surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness of single-use flexible ureteroscopes | 4 weeks postoperatively
  Comparison of total procedural cost and stone-free rate among three single-use flexible ureteroscopes used in retrograde intrarenal surgery (RIRS).

SECONDARY OUTCOMES:
Operative Time and Postoperative Complications | up to 4 weeks postoperatively
  Incidence of postoperative complications within the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham E Khayrallah, Resident, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No